CLINICAL TRIAL: NCT07405346
Title: Clinical Study on First-line Treatment for Advanced Leiomyosarcoma Based on Drug Sensitivity of Organoid
Brief Title: A Trial for Advanced Leiomyosarcoma With Human Organoid-guided Personalized Efficacy
Acronym: LMS-HOPE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Fudan University (Other); Zhejiang Cancer Hospital (Other); West China Hospital (Other); Xiangya Hospital of Central South University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Peking University Cancer Hospital & Institute (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); First Affiliated Hospital of Guangxi Medical University (Other); Hubei Cancer Hospital (Other); Henan Cancer Hospital (Other Government); Second Xiangya Hospital of Central South University (Other); Tianjin Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMS-HOPE
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Advanced Leiomyosarcoma
Keywords: Advanced Leiomyosarcoma; organoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group relying on organoid drug sensitivity results (Experimental): During the waiting period for organoid culture and drug sensitivity analysis results (approximately 3-4 weeks), all patients received one cycle of standard AI regimen chemotherapy (doxorubicin at least 50 mg/m ²+ifosfamide at least 6000 mg/m ²).
  Based on the results of drug sensitivity analysis and the patient's clinical response, comprehensively evaluate and adjust the treatment plan.
  Interventions: Drug: treatment based on the results of drug sensitivity analysis

INTERVENTIONS:
Drug: treatment based on the results of drug sensitivity analysis — During the waiting period for organoid culture and drug sensitivity analysis results (approximately 3-4 weeks), all patients received one cycle of standard AI regimen chemotherapy (doxorubicin at least 50 mg/m ²+ifosfamide at least 6000 mg/m ²).
  Based on the results of drug sensitivity analysis and the patient's clinical response, comprehensively evaluate and adjust the treatment plan.

SUMMARY:
This study is a prospective single arm multicenter intervention study aimed at evaluating the feasibility of using organoid drug sensitivity results to guide first-line treatment of advanced leiomyosarcoma. The primary endpoint of the study is objective response rate (ORR). The secondary endpoint are Progression Free Survival (PFS) and 6-month PFS rate.

DETAILED DESCRIPTION:
In this study, fresh tissues of the patient's primary lesion and/or metastatic lesion were obtained for constructing a tumor organoid model. Perform drug sensitivity analysis on the constructed organoids. During the waiting period for organoid culture and drug sensitivity analysis results (approximately 3-4 weeks), all patients received one cycle of standard AI regimen chemotherapy (doxorubicin at least 50 mg/m ²+ifosfamide at least 6000 mg/m ²).

Based on the results of drug sensitivity analysis and the patient's clinical response, comprehensively evaluate and adjust the treatment plan. By observing the clinical improvement status of patients, evaluate the accuracy and effectiveness of predicting drug efficacy based on organoid drug sensitivity results.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 75 years old, gender not limited;<p>
2. Patients pathologically confirmed leiomyosarcoma, who have not received systemic treatment in the advanced stage;<p>
3. According to the RECIST 1.1 standard, there are measurable target lesions present;<p>
4. The metastatic or primary lesion can obtain sufficient biopsy tissue;<p>
5. Eastern Cooperative Oncology Group (ECOG) performance status score ranges from 0 to 1, and for amputees, it can be relaxed to 2 points;<p>
6. Expected survival period ≥ 6 months;<p>
7. Good bone marrow reserve function: HB ≥ 90g/L; ANC≥1.5×109/L；PLT≥80×109/L；<p>
8. Good liver and kidney function reserve: BILS ≤ 1.5 times the upper limit of normal (ULN); ALT and AST ≤ 2.5 times ULN; Serum creatinine ≤ ULN;<p>
9. Good coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN, activated partial thromboplastin time (APTT) ≤ 1.5 times ULN;<p>
10. Female subjects with fertility must undergo a serum pregnancy test within 3 days before the first medication and the result must be negative. If a female subject with fertility has sexual intercourse with an unsterilized male partner, the subject must self screen and adopt an acceptable contraceptive method, and must agree to continue using the contraceptive method for 6 months after the last administration of the study drug; Whether to stop contraception after this point in time should be discussed with the researchers.<p>
11. The patient voluntarily joined this study and signed an informed consent form (ICF), with good compliance and cooperation with follow-up.

Exclusion Criteria:

1. Patients with peripheral nervous system disorders caused by diseases or those with a history of significant mental and central nervous system disorders;<p>
2. Patients with severe infections or active digestive ulcers requiring treatment;<p>
3. Those who are allergic to relevant therapeutic drugs or have surgical contraindications;<p>
4. Patients with other malignant tumors within the past 5 years, except for cured skin basal cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma, and other malignant tumors;<p>
5. Those whose heart function meets any of the following criteria: 1) Left ventricular ejection fraction (LVEF)<50% (detected by echocardiography). 2) The New York Heart Association (NYHA) has a heart function classification of ≥ II. 3) Clinically significant arrhythmias require drug treatment. 4) An acute myocardial infarction occurred within the 6 months prior to enrollment. 5) Uncontrolled hypertension (systolic blood pressure>160 mmHg or diastolic blood pressure>100 mmHg). 6) Other heart diseases that have been determined by researchers to be unsuitable for treatment with anthracyclines.<p>
6. Severe liver disease (such as cirrhosis), kidney disease, respiratory disease, blood system disease or uncontrollable diabetes;<p>
7. There are patients infected with hepatitis B, hepatitis C, syphilis and AIDS;<p>
8. Patients who relapse within 6 months after adjuvant chemotherapy;<p>
9. During the adjuvant therapy period, the cumulative equivalent dose of doxorubicin is greater than 120mg/m2;<p>
10. Patients who are currently participating or have participated in other clinical trials within the past month;<p>
11. Patients deemed unsuitable for inclusion by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | from the first drug administration up to two years
  ORR is the proportion of patients with best response of complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and iRECIST.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of first documented tumor progression or death due to any cause, whichever occurs first.
6-month PFS rate | from the first drug administration up to six month
  The proportion of patients who are still in a progression free survival state from the first systemic treatment to the total number of patients in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No